CLINICAL TRIAL: NCT02253342
Title: A Phase 1, Multiple-Dose, Open-Label Study to Determine and Compare Plasma and Intrapulmonary Pharmacokinetics of WCK 2349 in Healthy Adult Human Subjects
Brief Title: Study to Determine and Compare Plasma and Intrapulmonary Pharmacokinetics of WCK 2349 in Healthy Adult Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Clinartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: W-2349-103
Record Dates: First submitted 2014-09-23; First posted 2014-10-01 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Intrapulmonary Pharmacokinetics of WCK 2349

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WCK 2349 (Experimental): Subjects will receive oral doses of WCK 2349 administered twice-daily for five days starting on Day 1
  Interventions: Drug: WCK-2349

INTERVENTIONS:
Drug: WCK-2349 — Each subject will receive ten oral doses of 1000 mg WCK 2349 administered twice-daily starting on Day 1

SUMMARY:
This study to determine and compare plasma, epithelial lining fluid (ELF) and alveolar macrophage (AM) concentrations of levonadifloxacin after administration of WCK 2349 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females, 18 to 55 years of age (both inclusive) at the time of screening.
* Medical history without any major pathology as judged by the Principal Investigator.

Exclusion Criteria:

* History or presence of significant oncologic, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* Positive urine drug/alcohol testing at screening or confinement.
* Positive testing for HIV, Hepatitis B or Hepatitis C.
* History or presence of alcohol or drug abuse within the 2 years prior to screening.
* Excessive intake of alcohol, defined as an average daily intake of greater than three units, or an average weekly intake of greater than 21 units (one unit is equivalent to 1 can or bottle (12 oz) of beer, or 1 measure (1.5 oz) of spirits, or 1 glass (5 oz) of wine) in the last 6 months prior to screening.
* Known hypersensitivity to quinolones/fluoroquinolones.
* History of allergic or other serious adverse reactions to benzodiazepines or lidocaine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Concentrations of levonadifloxacin in WCK 2349 Epithelial lining fluid (ELF) and alveolar macrophage (AM) | 5 days
  Determine and compare plasma, epithelial lining fluid (ELF) and alveolar macrophage (AM) concentrations of levonadifloxacin after administration of WCK 2349

SECONDARY OUTCOMES:
Steady-state plasma pharmacokinetics of levonadifloxacin | 5 days
  To compare the steady-state plasma pharmacokinetics of levonadifloxacin following administration of WCK 2349
Safety and tolerability parameters-number of adverse event , change in clinical laboratory tests, ECG readings, change in physical examination and vital sign | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Gotfried, MD, Principal Investigator — Pulmonary Associates, PA
Locations (1):
- Pulmonary Associates, 1112 E. McDowell Rd., Phoenix, Arizona, United States

REFERENCES:
- [Derived] Rodvold KA, Gotfried MH, Chugh R, Gupta M, Yeole R, Patel A, Bhatia A. Intrapulmonary Pharmacokinetics of Levonadifloxacin following Oral Administration of Alalevonadifloxacin to Healthy Adult Subjects. Antimicrob Agents Chemother. 2018 Feb 23;62(3):e02297-17. doi: 10.1128/AAC.02297-17. Print 2018 Mar. PMID 29263070